CLINICAL TRIAL: NCT04344912
Title: Impact of COVID19 Outbreak in Cardiac Patients Admitted in Intensive Care Unit : the CCU-COVID19 Study
Brief Title: Impact of COVID19 Outbreak in Cardiac Acute Care
Acronym: CCU-COVID19
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Action, France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200524; 0522070420 (Other: INDS)
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acute Coronary Syndrome; Heart Failure; COVID
Keywords: COVID19; Acute Coronary Syndrome; Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure; COVID-19; Myocardial Infarction | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID19- Population: Patients without diagnosis of COVID19, as assessed by RT-PCR and CT scan
  Interventions: Other: Data collection
- COVID19+ Population: Patients with a diagnosis of COVID19, as assessed by RT-PCR and CT scan
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Diagnostic and prognostic evaluation of cardiac patients hospitalized in CCU during the COVID-19 outbreak; patient's immune status regarding the presence of SARS-CoV-2 specific antibodies

SUMMARY:
This registry will evaluate the impact of the COVID19 outbreak on Cardiac patients admitted in the Intensive Care Unit of the Pitie-Salpetriere Hospital in Paris, France

DETAILED DESCRIPTION:
Registry on Characteristics and outcomes of Cardiac patients (COVID- and COVID+) hospitalized in the Intensive Care Unit of the Pitie-Salpetriere Hospital in Paris, France

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Admitted in the Cardiac Intensive Care Unit from March 20th 2020
* Patient informed and having expressed his non-opposition to participate in the research

Exclusion Criteria:

* Minor patient
* Patient who expressed opposition to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated in the CCU at Cardiology Institute of the Pitié-Salpêtrière Hospital, from Friday, March 20, 2020
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of recurrent Major Cardiovascular Events (MACE) and urgent rehospitalization | From admission to one year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Johanne SILVAIN, MD PhD, Study Director — Sorbonne University, ACTION Group, AP-HP Pitié-Salpêtrière Hospital Paris France; Gilles MONTALESCOT, MD PhD, Study Chair — Sorbonne University, ACTION Group, AP-HP Pitié-Salpêtrière Hospital Paris France
Locations (1):
- Unité de Soins Intensifs de Cardiologie, Pitié Salpêtrière Hospital, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Open to collaboration
Time Frame: The data will be available 12 months after the beginning of the Registry
Access Criteria: to be determined